CLINICAL TRIAL: NCT03829254
Title: A Phase I/II, Open-label, Dose-escalation and Expansion Study to Assess the Safety, Pharmacokinetics and Clinical Activity of NUC-7738, a Nucleotide Analogue, in Patients With Advanced Solid Tumours and Lymphoma
Brief Title: A Safety, Pharmacokinetic and Clinical Activity Study of NUC-7738 in Patients With Advanced Solid Tumours and Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NuCana plc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NuTide:701; 2018-003417-17 (EudraCT Number)
Record Dates: First submitted 2019-01-30; First posted 2019-02-04 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Cancer; Lymphoma; Solid Tumor; Melanoma
Keywords: Solid tumors; Lymphoma; Cordycepin; Pembrolizumab; Melanoma
MeSH Terms: conditions — Lymphoma; Melanoma | interventions — NUC-7738; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NUC-7738 (Experimental): NUC-7738 administered by intravenous infusion on a weekly or fortnightly schedule. In the weekly dosing schedule, NUC-7738 is administered on Days 1 and 8 of a 14-day cycle. In the fortnightly dosing schedule, NUC-7738 is administered on Day 1 of a 14-day cycle.
  Interventions: Drug: NUC-7738
- NUC-7738 + pembrolizumab (Experimental): NUC-7738 administered by intravenous infusion on a weekly schedule on Days 1, 8 and 15 of a 21-day cycle. Pembrolizumab administered by intravenous infusion every 3 weeks on Day 1 of a 21-day cycle.
  Interventions: Drug: NUC-7738; Drug: Pembrolizumab

INTERVENTIONS:
Drug: NUC-7738 — NUC-7738
  Other Names: Nucleotide Analogue
Drug: Pembrolizumab — Pembrolizumab
  Other Names: Keytruda
  Arms: NUC-7738 + pembrolizumab

SUMMARY:
This is a Phase I/II, dose-escalation and expansion study of NUC-7738 administered by intravenous infusion as a monotherapy and in combination with pembrolizumab.

In Phase I, NUC-7738 monotherapy is evaluated across two administration schedules (weekly or fortnightly) in a dose-escalation design in patients with advanced solid tumours. The main objectives are to assess the safety and tolerability of NUC-7738, in addition to establishing the Maximum Tolerated Dose (MTD) and dose administration schedule of NUC-7738 for further exploration in the Phase II part of the study.

In Phase II, the selected dose and designated dosing schedule will be further evaluated in dose-confirmation expansion cohorts enrolling a total of approximately 40 additional patients with advanced solid tumours. Based on emerging data, approximately 6 patients with cutaneous melanoma will be enrolled to these expansion cohorts and will receive NUC-7738 monotherapy. A further cohort will assess NUC-7738 in combination with pembrolizumab in approximately 6-12 patients with cutaneous melanoma. Based on efficacy signals observed in the initial melanoma combination cohort, a further expansion cohort will be initiated to expand to a total of 40 patients to allow a powered analysis. In addition, 12 patients with lymphoma (with potential expansion to a total of 25 patients) may be enrolled to receive NUC-7738 monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed written informed consent.
2. Solid tumour cohorts only (Phase I and Phase II; excluding NUC-7738 + pembrolizumab cohort): Histologically confirmed diagnosis of an advanced solid tumour with measurable disease as per RECIST v1.1 criteria and/or evaluable disease (evaluable: cytologically or radiologically detectable disease such as ascites, peritoneal deposits, or lesions, which do not fulfil RECIST v1.1 criteria for measurable disease) for solid tumours.
3. NUC-7738 + pembrolizumab cohort only (Phase II): Histologically confirmed diagnosis of metastatic cutaneous melanoma with measurable disease as per RECIST v1.1 criteria. Must have progressed on ≤2 prior lines of therapy for advanced/metastatic disease. In addition, patients may have been treated in the neoadjuvant/adjuvant setting. At least one prior line must have included a PD-1/PD-L1-containing regimen (either monotherapy or in combination) for which they progressed on.
4. Lymphoma cohort only (Phase II): Relapsed refractory lymphoma (high grade and low grade B-NHL, Hodgkin's Lymphoma and T-cell lymphomas), which is not amenable to standard of care, is refractory to standard of care or for which no standard of care exists. Patients must have bi-dimensionally measurable disease as per Cheson et al, 2007 criteria for lymphoma.
5. For solid tumours in single-agent Phase II cohorts only: patients should have received no more than 3 prior lines of treatment for metastatic disease.
6. Age ≥18 years (no upper age limit).
7. Eastern Cooperative Oncology Group performance status of 0 or 1.
8. Life expectancy of ≥12 weeks.
9. Adequate bone marrow, liver, and renal function.
10. Ability to comply with protocol requirements.
11. Female patients of child-bearing potential must have a negative serum pregnancy test within 3 days prior to the first NUC-7738 administration. All patients of child-bearing potential must agree to practice true abstinence or to use two forms of contraception, one of which must be a highly effective method of contraception, from the time of screening until 6 months after the last dose of study medication.
12. Phase I and Phase II dose-confirmation cohorts only: Patient must be willing to undergo a new tumour biopsy at Screening and during therapy on the study. Biopsies are mandatory for patient inclusion, except where taking a biopsy would be associated with unacceptable clinical risk due to the location of the disease. Such patients may be discussed on a case-by-case basis with the study Medical Monitor to determine their eligibility. A prior (archival) biopsy that is less than 3 months old may be substituted for a fresh tumour biopsy at Screening with agreement from the Medical Monitor. From protocol v3.4 onwards, biopsies are no longer required.
13. Patients must have been advised to take measures to avoid or minimise exposure of the skin and eyes to UV light, including avoiding sunbathing and visits to the solarium, for the duration of study participation and for a period of 4 weeks following the last dose of study medication.

Exclusion Criteria:

The following exclusion criteria apply to all patients. Please also refer to additional exclusion criteria for the NUC-7738 + pembrolizumab cohort below.

1. History of allergic reaction fo any of the components of NUC-7738.
2. Central nervous system or leptomeningeal metastases. Patients with brain metastases are eligible if they have no ongoing neurological symptoms, have not received corticosteroids within 7 days prior to enrolment, and show radiographic stability for at least 2 weeks.
3. Chemotherapy, radiotherapy (other than a short cycle of palliative radiotherapy for bone pain), immunotherapy, or exposure to another investigational agent within 28 days (for biological agents decision on washout period will be made on a case by base basis) of first administration of the IMP:

   1. For nitrosoureas and mitomycin C within 6 weeks of first administration of NUC-7738
   2. For hormone therapy within 14 days of first administration of NUC-7738
   3. Corticosteroid treatment is allowed during the screening period but should be weaned to a dose of 10 mg prednisolone (or steroids equivalent) by Cycle 1 Day 1.
4. Prior toxicities from anti-cancer agents or radiotherapy, which have not regressed to Grade ≤1 severity (NCI-CTCAE v5.0), excluding neuropathy, ototoxicity and alopecia (which are excluded if ≥Grade 3).
5. Presence of any uncontrolled concomitant illness, serious illness, medical conditions, or other medical history, including laboratory results, which, in the Investigator's opinion, would be likely to interfere with their participation in the study, or with the interpretation of results, including the following:

   1. Congestive heart failure (New York Heart Association Class III or Class IV).
   2. Myocardial infarction within 6 months of the first dose of study medication.
   3. Unstable or poorly controlled angina pectoris.
   4. Complete left bundle branch, bifascicular block or other clinically significant abnormal electrocardiogram finding.
   5. A history of or current risk factor for Torsades de Point (e.g., heart failure, hypokalaemia, or a family history of long QT syndrome).
   6. A history of, or current diagnosis of, interstitial pneumonitis or pulmonary fibrosis.
6. Known human immunodeficiency virus positive or known active hepatitis B or C. Presence of an active bacterial or viral infection including Herpes zoster or chicken pox.
7. Any condition (e.g., known or suspected poor compliance, psychological instability, geographical location etc.) that, in the judgment of the Investigator, may affect the patient's ability to sign the informed consent and undergo study procedures.
8. Currently pregnant, lactating or breastfeeding.
9. QTc interval >450 milliseconds for males and >470 milliseconds for females.
10. Concomitant use of drugs known to prolong QT/QTc interval.
11. Concomitant use of strong CYP3A4 inducers or strong CYP3A4 inhibitors. The use of strong CYP3A4 inducers within 2 weeks of first receipt of study drug or the use of strong CYP3A4 inhibitors within 1 week of first receipt of study drug is also excluded.
12. Have received a live vaccination within four weeks of first planned dose of study medication.

NUC-7738 + pembrolizumab cohort only

1. Any history of hypersensitivity or current contra-indication to the components of pembrolizumab (L-histidine, polysorbate 80, sucrose, sodium hydroxide, hydrochloric acid).
2. Current contra-indication to immunotherapy with checkpoint inhibitors.
3. Systemic steroid therapy or any immunosuppressive therapy (≥10 mg/day prednisone or equivalent).
4. Known neutralising antibodies against checkpoint inhibitors.
5. Patients previously exposed to checkpoint inhibitors who are not adequately treated for skin rash or have no replacement therapy for endocrinopathies.
6. Any prior toxicity attributed to checkpoint inhibitors that resulted in discontinuation of therapy. These patients should be discussed on a case-by-case basis with the Medical Monitor.
7. Active autoimmune disease or a documented history of autoimmune disease, including ulcerative colitis and Crohn's disease or any condition that requires systemic steroids.
8. Prior treatment with cell therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicities | From the date of consent until 30 days after the last dose of NUC-7738 administered
  Phase I: Safety and tolerability of NUC-7738 in patients with advanced solid tumours
Number of patients with treatment-emergent adverse events (CTCAE v5.0) | From the date of consent until 30 days after the last dose of NUC-7738 administered
  Phase I: Safety and tolerability of NUC-7738 in patients with advanced solid tumours
Number of patients with clinically significant laboratory changes (CTCAE v5.0) | From the date of consent until 30 days after the last dose of NUC-7738 administered
  Phase I: Safety and tolerability of NUC-7738 in patients with advanced solid tumours
Number of patients with changes in physical exam, vital signs, and serial electrocardiograms. | From the date of consent until 30 days after the last dose of NUC-7738 administered
  Phase I: Safety and tolerability of NUC-7738 in patients with advanced solid tumours
MTD for NUC-7738 administered via weekly and fortnightly dosing schedules in patients with advanced solid tumours | Until completion of Phase I (an average of 1 year)
  Phase I
Percentage change from baseline in tumour size | Assessed every 8 weeks following Day 1 up to and including Cycle 12 (each cycle is 14 days) in single-agent cohorts and Cycle 8 in combination cohorts (each cycle is 21 days), moving to every 12 weeks until the end of study (up to 22 months)
  Phase II: Efficacy (per RECIST v 1.1, iRECIST or Cheson et al, 2007)
Objective response rate (ORR) | Assessed every 8 weeks following Day 1 up to and including Cycle 12 (each cycle is 14 days) in single-agent cohorts and Cycle 8 in combination cohorts (each cycle is 21 days), moving to every 12 weeks until the end of study (up to 22 months)
  Phase II: Efficacy (per RECIST v 1.1, iRECIST or Cheson et al, 2007): defined as the number of patients achieving a confirmed response (complete response [CR] or partial response [PR])
Duration of response (DoR) | Assessed every 8 weeks following Day 1 up to and including Cycle 12 (each cycle is 14 days) in single-agent cohorts and Cycle 8 in combination cohorts (each cycle is 21 days), moving to every 12 weeks until the end of study (up to 22 months)
  Phase II: Efficacy (per RECIST v 1.1, iRECIST or Cheson et al, 2007): defined as the time from the time measurement criteria are first met for CR or PR until the first date that recurrence or progressive disease (PD) is objectively documented (responders only)
Disease control rate (DCR) | Assessed every 8 weeks following Day 1 up to and including Cycle 12 (each cycle is 14 days) in single-agent cohorts and Cycle 8 in combination cohorts (each cycle is 21 days), moving to every 12 weeks until the end of study (up to 22 months)
  Phase II: Efficacy (per RECIST v 1.1, iRECIST or Cheson et al, 2007): defined as the proportion of patients achieving confirmed response (CR and PR) or stable disease (SD) as the best overall response
Duration of stable disease (DoSD) | Assessed every 8 weeks following Day 1 up to and including Cycle 12 (each cycle is 14 days) in single-agent cohorts and Cycle 8 in combination cohorts (each cycle is 21 days), moving to every 12 weeks until the end of study (up to 22 months)
  Phase II: Efficacy (per RECIST v 1.1, iRECIST or Cheson et al, 2007): defined as the time from the time measurement criteria are first met for SD until the first date that recurrence or PD is objectively documented
Progression free survival (PFS) | Assessed every 8 weeks following Day 1 up to and including Cycle 12 (each cycle is 14 days) in single-agent cohorts and Cycle 8 in combination cohorts (each cycle is 21 days), moving to every 12 weeks until the end of study (up to 22 months)
  Phase II: Efficacy (per RECIST v 1.1, iRECIST or Cheson et al, 2007): defined as the time from first dose of study treatment until the date of objective disease progression or death

SECONDARY OUTCOMES:
Phase I: Plasma concentration of NUC-7738 at end of infusion (Cinf) | Samples collected on Days 1, 2, and 3 of Cycle 1 and Days 1 and 2 of Cycle 2 (cycle: 14 days).
Phase I: Maximum observed plasma concentration (Cmax) of NUC-7738, 3'-dA, 3'-deoxyinosine (3'-dI) and alanine phosphate metabolite of NUC-7738 | Samples collected on Days 1, 2, and 3 of Cycle 1 and Days 1 and 2 of Cycle 2 (cycle: 14 days).
Phase I: Area under the plasma concentration-time curve (AUC) of NUC-7738, 3'-dA, 3'-deoxyinosine (3'-dI) and alanine phosphate metabolite of NUC-7738 | Samples collected on Days 1, 2, and 3 of Cycle 1 and Days 1 and 2 of Cycle 2 (cycle: 14 days).
Phase I: Elimination half-life (t½) of NUC-7738, 3'-dA, 3'-deoxyinosine (3'-dI) and alanine phosphate metabolite of NUC-7738 | Single-agent cohorts: Samples collected on Days 1, 2 and 3 of each dose level (cycle: 14 days). Combination cohorts: Samples collected on Days 1, 2, and 3 of Cycle 1 and on Day 1 of the dose escalation step (cycle: 21 days)
Phase I: Volume of distribution of NUC-7738, 3'-dA, 3'-deoxyinosine (3'-dI) and alanine phosphate metabolite of NUC-7738 | Single-agent cohorts: Samples collected on Days 1, 2 and 3 of each dose level (cycle: 14 days). Combination cohorts: Samples collected on Days 1, 2, and 3 of Cycle 1 and on Day 1 of the dose escalation step (cycle: 21 days)
Phase I: Clearance of NUC-7738, 3'-dA, 3'-deoxyinosine (3'-dI) and alanine phosphate metabolite of NUC-7738 | Single-agent cohorts: Samples collected on Days 1, 2 and 3 of each dose level (cycle: 14 days). Combination cohorts: Samples collected on Days 1, 2, and 3 of Cycle 1 and on Day 1 of the dose escalation step (cycle: 21 days)
Phase II: Plasma concentration of NUC-7738 at end of infusion (Cinf) | Single-agent cohorts: Samples collected on Days 1, 2 and 3 of each dose level (cycle: 14 days). Combination cohorts: Samples collected on Days 1, 2, and 3 of Cycle 1 and on Day 1 of the dose escalation step (cycle: 21 days)
Phase II: Maximum observed plasma concentration (Cmax) of NUC-7738, 3'-dA, 3'-deoxyinosine (3'-dI) and alanine phosphate metabolite of NUC-7738 | Single-agent cohorts: Samples collected on Days 1, 2 and 3 of each dose level (cycle: 14 days). Combination cohorts: Samples collected on Days 1, 2, and 3 of Cycle 1 and on Day 1 of the dose escalation step (cycle: 21 days)
Phase II: Area under the plasma concentration-time curve (AUC) of NUC-7738, 3'-dA, 3'-deoxyinosine (3'-dI) and alanine phosphate metabolite of NUC-7738 | Single-agent cohorts: Samples collected on Days 1, 2 and 3 of each dose level (cycle: 14 days). Combination cohorts: Samples collected on Days 1, 2, and 3 of Cycle 1 and on Day 1 of the dose escalation step (cycle: 21 days)
Phase II: Elimination half-life (t½) of NUC-7738, 3'-dA, 3'-deoxyinosine (3'-dI) and alanine phosphate metabolite of NUC-7738 | Single-agent cohorts: Samples collected on Days 1, 2 and 3 of each dose level (cycle: 14 days). Combination cohorts: Samples collected on Days 1, 2, and 3 of Cycle 1 and on Day 1 of the dose escalation step (cycle: 21 days)
Phase II: Volume of distribution of NUC-7738, 3'-dA, 3'-deoxyinosine (3'-dI) and alanine phosphate metabolite of NUC-7738 | Single-agent cohorts: Samples collected on Days 1, 2 and 3 of each dose level (cycle: 14 days). Combination cohorts: Samples collected on Days 1, 2, and 3 of Cycle 1 and on Day 1 of the dose escalation step (cycle: 21 days)
Phase II: Clearance of NUC-7738, 3'-dA, 3'-deoxyinosine (3'-dI) and alanine phosphate metabolite of NUC-7738 | Single-agent cohorts: Samples collected on Days 1, 2 and 3 of each dose level (cycle: 14 days). Combination cohorts: Samples collected on Days 1, 2, and 3 of Cycle 1 and on Day 1 of the dose escalation step (cycle: 21 days)
Percentage change from baseline in tumour size | Assessed every 8 weeks following Day 1 up to and including Cycle 12 (each cycle is 14 days), moving to every 12 weeks until the end of study (up to 22 months)
  Phase I: Efficacy (per RECIST v 1.1 or Cheson et al, 2007)
  The percentage change in the sum of longest diameters of target lesions from baseline to Week 8.
  The best percentage change in the sum of longest diameters of target lesions from baseline to best on-treatment measurement
ORR | Assessed every 8 weeks following Day 1 up to and including Cycle 12 (each cycle is 14 days), moving to every 12 weeks until the end of study (up to 22 months)
  Phase I: Efficacy (per RECIST v 1.1 or Cheson et al, 2007): defined as the number of patients achieving a confirmed response (complete response [CR] or partial response [PR])
DoR | Assessed every 8 weeks following Day 1 up to and including Cycle 12 (each cycle is 14 days), moving to every 12 weeks until the end of study (up to 22 months)
  Phase I: Efficacy (per RECIST v 1.1 or Cheson et al, 2007): defined as the time from the time measurement criteria are first met for CR or PR until the first date that recurrence or progressive disease (PD) is objectively documented (responders only)
DCR | Assessed every 8 weeks following Day 1 up to and including Cycle 12 (each cycle is 14 days), moving to every 12 weeks until the end of study (up to 22 months)
  Phase I: Efficacy (per RECIST v 1.1 or Cheson et al, 2007): defined as the proportion of patients achieving confirmed response (CR and PR) or stable disease (SD) as the best overall response
DoSD | Assessed every 8 weeks following Day 1 up to and including Cycle 12 (each cycle is 14 days), moving to every 12 weeks until the end of study (up to 22 months)
  Phase I: Efficacy (per RECIST v 1.1 or Cheson et al, 2007): defined as the time from the time measurement criteria are first met for SD until the first date that recurrence or PD is objectively documented
PFS | Assessed every 8 weeks following Day 1 up to and including Cycle 12 (each cycle is 14 days), moving to every 12 weeks until the end of study (up to 22 months)
  Phase I: Efficacy (per RECIST v 1.1 or Cheson et al, 2007): defined as the time from first dose of study treatment until the date of objective disease progression or death
Number of patients with treatment-emergent adverse events (CTCAE v5.0) | From the date of consent until 30 days after the last dose of NUC-7738 administered
  Phase II: Safety and tolerability of NUC-7738 as a single-agent or in combination with pembrolizumab in patients with advanced solid tumours and lymphoma
Number of patients with clinically significant laboratory changes (CTCAE v5.0) | From the date of consent until 30 days after the last dose of NUC-7738 administered
  Phase II: Safety and tolerability of NUC-7738 as a single-agent or in combination with pembrolizumab in patients with advanced solid tumours and lymphoma
Number of patients with changes in physical exam, vital signs, and serial electrocardiograms. | From the date of consent until 30 days after the last dose of NUC-7738 administered
  Phase II: Safety and tolerability of NUC-7738 as a single-agent or in combination with pembrolizumab in patients with advanced solid tumours and lymphoma

CONTACTS AND LOCATIONS:
Locations (9):
- United Kingdom (9):
  - Cambridge University Hospitals NHS Foundation Trust (Addenbrookes Hospital), Cambridge
  - Edinburgh Cancer Centre, Western General Hospital, Edinburgh
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - University College London Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Freeman Hospital, Newcastle
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Lancashire Teaching Hospitals NHS Foundation Trust, Royal Preston Hospital, Preston

IPD SHARING:
Plan to Share IPD: No